CLINICAL TRIAL: NCT06561113
Title: Does a Cup of Turkish Coffee Affect Postural Control and Hand-eye Coordination in Young Adults? A Quasi-experimental Study
Brief Title: The Effect of Turkish Coffee on Postural Control and Hand-eye Coordination in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Deniz Tuncer, Asst. Prof. Deniz Tuncer, Bezmialem Vakif University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 29.07.2024-159880
Record Dates: First submitted 2024-08-13; First posted 2024-08-19 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Caffeine; Balance; Distorted; Coordination and Balance Disturbances

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Participants who meet the inclusion and exclusion criteria will undergo postural control assessment with the Biodex Balance System® and hand-eye coordination test with the Alternate Hand Wall Toss Test. Subjects will be given 65 ml of Turkish coffee (one cup) to ensure oral caffeine intake. The same assessments will be repeated 30 minutes after caffeine intake.
  Interventions: Other: Caffeine intake

INTERVENTIONS:
Other: Caffeine intake — One cup of Turkish coffee contains 60 mg/65 ml (1 Turkish coffee cup) of caffeine. Participants will be instructed to sit for 10 minutes before drinking coffee. To prepare the Turkish coffee, 5 g of ground dry coffee will be mixed in 100 mL of tap water and left to boil in a coffee machine. When the first boil starts, it will be removed from the machine and poured into the cup. Then, 65 ml of Turkish coffee will be given to the subjects to ensure oral caffeine intake.

SUMMARY:
Although the effects of different doses of caffeine on balance have been evaluated in various studies, the effects of low doses of caffeine ingested with Turkish coffee on postural control and hand-eye coordination remain unclear. In this study, it will be investigated the acute effects of 60 mg caffeine intake via Turkish coffee on postural control and hand-eye coordination.

DETAILED DESCRIPTION:
This study is designed as a one-group pretest-posttest quasi-experimental research. The study will be conducted with healthy young adults with low coffee consumption habits. Participants who meet the inclusion and exclusion criteria will undergo postural control assessment with the Biodex Balance System® and hand-eye coordination test with the Alternate Hand Wall Toss Test. Subjects will be given 65 ml of Turkish coffee (one cup) to ensure oral caffeine intake. The same assessments will be repeated 30 minutes after caffeine intake.

ELIGIBILITY:
Inclusion Criteria:

* Being 18-26 years of age
* Having a normal body mass index

Exclusion Criteria:

* Having a health problem that prevented caffeine intake
* Having a diagnosis of vestibular and neurological disease
* Using drugs that affect the central nervous system
* Using any medication related to chronic disease
* Having lower extremity rotational alignment disorder
* Having a history of lower and/or upper extremity injury or surgery in the last year

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-08-14 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
Postural control assessment with Biodex Balance System | Baseline and immediately after caffeine intake
  Postural control evaluation will be performed with "Biodex Balance System" (Shirley, NY). Three tests will be performed with the device: postural stability test, stability limits test, and the Modified Clinical Test for Sensory Interaction and Balance (mCTSIB). The test will then continue for 30 seconds, during which time the number of balls caught will be noted

SECONDARY OUTCOMES:
Hand-eye coordination assessment with alternate hand-wall toss test | Baseline and immediately after caffeine intake
  Alternate hand wall toss test will be used to measure hand-eye coordination. The Alternate-Hand Wall-Toss Test is a test of hand-eye coordination, where the participant throw a ball against a wall from one hand in an underarm action, and attempt to catch it with the opposite hand. The test will then continue for 30 seconds, during which time the number of balls caught will be noted.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided